CLINICAL TRIAL: NCT07210047
Title: A Phase Ib/II Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Efficacy of HuL001 in Combination With Lenalidomide and Dexamethasone in Subjects With Relapsed/Refractory Multiple Myeloma
Brief Title: Study of HuL001 in Relapsed/Refractory Multiple Myeloma Patients
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: HuniLife Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HuL001-CT-102
Record Dates: First submitted 2025-09-19; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma Refractory
Keywords: Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose escalation Cohort 1 (Active Comparator): HuL001, Lenalidomide and Dexamethasone
  Interventions: Biological: HuL001-10 mg/kg; Drug: Lenalidomide and Dexamethasone
- Dose escalation Cohort 2 (Active Comparator): HuL001, Lenalidomide and Dexamethasone
  Interventions: Biological: HuL001-15 mg/kg; Drug: Lenalidomide and Dexamethasone
- Dose expansion Cohort 3 (Active Comparator): HuL001, Lenalidomide and Dexamethasone
  Interventions: Biological: HuL001-10 mg/kg; Biological: HuL001-15 mg/kg; Drug: Lenalidomide and Dexamethasone

INTERVENTIONS:
Biological: HuL001-10 mg/kg — Anti-ENO1 monoclonal antibody
  Other Names: Anti-ENO1 monoclonal antibody
  Arms: Dose escalation Cohort 1; Dose expansion Cohort 3
Biological: HuL001-15 mg/kg — Anti-ENO1 monoclonal antibody
  Arms: Dose escalation Cohort 2; Dose expansion Cohort 3
Drug: Lenalidomide and Dexamethasone — Lenalidomide in combination with dexamethasone is indicated for the treatment of adult patients with multiple myeloma (MM)

SUMMARY:
The goal of this clinical trial is to learn if the antibody drug HuL001, combined with

Lenalidomide/Dexamethasone works to treat Multiple Myeloma patients. It will also learn about the safety and tolerability of the therapeutic combination. The objectives of this study are:

1. To evaluate the safety and tolerability of HuL001 (in combination with Len/Dex).
2. To evaluate the efficacy of HuL001 (in combination with Len/Dex).

Researchers will use the antibody drug HuL001, combined with Len/Dex, to see if this works for Multiple Myeloma therapy.

Participants will:

* Receive HuL001 antibody injections every 2 weeks
* Take Lenalidomide for 21 consecutive days each month
* Take Dexamethasone every 1 week
* Visit the clinic on scheduled days for checkups and tests
* Keep a diary of their symptoms and Myeloma responses.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet ALL inclusion criteria will be included.

1. Subjects aged 18 (inclusive) or older.
2. Confirmed diagnosis of RRMM according to the IMWG guidelines (International Myeloma Working Group updated criteria for the diagnosis of multiple myeloma, 2016).
3. Subjects must have one or more of the following measurable disease criteria:

   1. Serum M-protein level ≥ 0.5 g/dL.
   2. Urine M-protein level ≥ 200 mg/24 hours.
   3. Light chain MM without measurable M-protein in the serum or urine: Serum immunoglobulin free light chain ≥ 10 mg/dL (local lab) and abnormal serum immunoglobulin kappa lambda free light chain ratio (per normal ranges of local lab).
4. Subjects have disease progression on, refractory to, or intolerant to at least 3 prior lines of anti-myeloma therapies or 2 prior lines of therapies with three different drugs, including an anti-CD38 monoclonal antibody, a proteasome inhibitor, and an immunomodulatory drug, and are refractory to at least one of these drugs, or who are unwilling to receive or ineligible for other standard therapies according to local medical practice.
5. There must be a time interval ≥ 3 months between the prior hematopoietic cell transplantation (HCT, counted as 1 prior line of therapy) and the first dose of HuL001.
6. All toxicities associated with the prior anti-myeloma therapy have recovered to Grade 1 or baseline at the screening.
7. Eastern Cooperative Oncology Group (ECOG) performance score of 0-1.
8. Life expectancy ≥ 6 months in the opinion of the investigator.
9. Adequate organ functions are defined as follows.

   1. Hemoglobin ≥ 8.5 g/dL.
   2. White blood cell (WBC) count ≥ 2.5 x 103/μL.
   3. Neutrophil count ≥ 1.5 × 103/μL.
   4. Platelet count ≥ 80 × 103/μL.
   5. Aspartate aminotransferase (AST) ≤ 2.5 × upper limit of normal (ULN).
   6. Alanine aminotransferase (ALT) ≤ 2.5 × ULN.
   7. Total bilirubin ≤ 2 × ULN.
   8. Creatinine clearance (CrCl) ≥ 60 mL/min, calculated using Cockcroft-Gault formula.

   Notes:
   1. Subjects receiving hematopoietic growth factor support, e.g., erythropoietin, granulocyte-colony stimulating factor, platelet stimulator, etc. must have a 2-week interval between growth factor support and the screening evaluation. They may receive growth factor support after the DLT assessment period during the study.
   2. There must be at least a 2-week interval between the last red blood cell (RBC) transfusion and hemoglobin assessment at the screening and at least a 1-week interval between the last platelet transfusion and the platelet assessment at the screening. Subjects may receive RBC and platelet transfusion after the DLT assessment period during the study.
10. Negative serology test for Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), and Hepatitis C Virus (HCV) infection. Note: If a subject with positive anti-HCV Ab, the subject must be with negative HCV RNA for enrollment. If a subject with positive HBsAg, the subject must be with undetectable HBV DNA for enrollment.
11. Female subject with reproductive potential must have a negative result of serum pregnancy test at the screening visit and urine pregnancy test before each cycle of HuL001 administration.
12. Female subject with reproductive potential and male subject with reproductive potential must agree to refrain from unprotected sex and use 2 methods of highly effective contraception with their partner (e.g., barrier contraceptives [male condom, female condom, or diaphragm plus spermicide], intrauterine device, hormonal methods [hormone shot or injection, implants, combination oral contraceptives, or patches]) for ≥ 6 months after the last dose of HuL001.
13. Physically and mentally capable of participating in the study and willing to adhere to study procedures.
14. Provision of signed informed consent.

Exclusion Criteria:

Subjects who meet ANY exclusion criteria will be excluded.

1. Suspected or known contraindication or intolerant reaction to lenalidomide and/or dexamethasone.
2. Suspected or known hypersensitivity (including allergy) to any of the components of the HuL001, lenalidomide, or dexamethasone.
3. Previous history of anaphylaxis and severe allergic reaction, generation of neutralizing antibodies, or hypersensitivity to albumin or a protein-based therapeutic, or any other mAb.
4. Planning to receive the HCT during the study period (approximately 6 months following the first dose of HuL001).
5. Active graft versus host diseases (GvHD) following the prior HCT.
6. Will be on digoxin therapy throughout the study period.
7. Presence of multiple primary cancers with the exception of carcinoma in situ and skin cancers after curative surgery.
8. Central nervous system (CNS) or meningeal involvement of MM by clinical signs or imaging studies.
9. Significant infections requiring systemic treatment within 1 month prior to the first dose of HuL001.
10. History of active tuberculosis in line with local medical practice.
11. Major surgery within 4 weeks prior to the first dose of HuL001. Subjects should be fully recovered from any surgically related complications.
12. Receipt of radiation therapy or systemic anti-MM treatments within 2 weeks prior to the first dose of HuL001.
13. Receipt of any live or live attenuated vaccine (e.g., varicella, pneumococcus) within 4 weeks prior to the first dose of HuL001 or planning to receive live vaccine during the study period. Seasonal flu and COVID-19 vaccines not containing live virus are permitted.
14. Any known active gastrointestinal dysfunction interfering with subject's ability to swallow tablets or any known active gastrointestinal dysfunction that could interfere with absorption of study drugs as judged by the investigator.
15. Myocardial infarction, unstable angina, or poorly controlled arrhythmia within 6 months prior to the screening visit.
16. Evidence or history of severe intercurrent medical conditions or clinically significant comorbidities that may interfere with optimal participation in the study or place the subject at increased risk of adverse events, including but not limited to psychiatric, ophthalmic, hematologic, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, immunologic, metabolic, urologic, dermatologic, neurologic, or allergic diseases, or other significant clinical findings within 3 months prior to the screening, as judged by the Investigator.
17. Receipt of any investigational drug or device or participation in a clinical study within 28 days prior to the V2(C1D1).
18. History of substance or alcohol abuse within 6 months prior to the screening visit.
19. Female subjects who are pregnant, breastfeeding, or planning to be pregnant or breastfeeding during the screening and study period.
20. Subject who is considered unfit to participate in the clinical study as assessed by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Myeloma responses | From enrollment to the end of treatment at 8 months
  Myeloma responses as assessed by the investigator according to the IMWG criteria

SECONDARY OUTCOMES:
Safety parameters | From enrollment to the end of treatment at 8 months
  Safety parameters as assessed by the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 during the study period.
PK parameter: Cmax | From enrollment to the end of treatment at 8 months
  PK parameter in the serum: Cmax
PK parameter: Tmax | From enrollment to the end of treatment at 8 months
  PK parameter in the serum: Tmax
PK parameter: AUCtau | From enrollment to the end of treatment at 8 months
  PK parameter in the serum: AUCtau
PK parameter: AUCinf | From enrollment to the end of treatment at 8 months
  PK parameter in the serum: AUCinf
PK parameter: t1/2 | From enrollment to the end of treatment at 8 months
  PK parameter in the serum: t1/2
Immunogenicity | From enrollment to the end of treatment at 8 months
  Immunogenicity: Anti-HuL001 antibodies (ADA).

CONTACTS AND LOCATIONS:
Overall Officials: Maisie Huang, PhD, Study Director — HuniLife Biotechnology
Locations (1):
- Far Eastern Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
There are no current plans to prepare IPD for sharing due to resource limitations.